CLINICAL TRIAL: NCT02389881
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Safety, Tolerability, and Pharmacokinetic Study in Healthy Subjects After Multiple Oral Doses of TAK-058
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple-Dose TAK-058 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-058-1002; U1111-1165-3644 (Other: WHO)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 Non-elderly Healthy: TAK-058 25 mg (Experimental): TAK-058 25 mg solution, orally, once daily on Day 1 and Days 4 through 10, in non-elderly healthy participants.
  Interventions: Drug: TAK-058
- Cohort 2 Non-elderly Healthy: TAK-058 75 mg (Experimental): TAK-058 75 mg solution, orally, once daily on Day 1 and Days 4 through 10, in non-elderly healthy participants.
  Interventions: Drug: TAK-058
- Cohort 3 Non-elderly Healthy: TAK-058 150 mg (Experimental): TAK-058 150 mg solution, orally, once daily on Day 1 and Days 4 through 10, in non-elderly healthy participants.
  Interventions: Drug: TAK-058
- Cohort 4 Elderly Healthy: TAK-058 25 mg (Experimental): TAK-058 25 mg solution, orally, once daily on Day 1 and Days 4 through 10, in elderly healthy participants.
  Interventions: Drug: TAK-058
- Cohort 5 Non-elderly Healthy: TAK-058 300 mg (Placebo Comparator): TAK-058 300 mg solution, orally, once daily on Day 1, in non-elderly healthy participants.
  Interventions: Drug: TAK-058
- Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo (Placebo Comparator): TAK-058 placebo-matching solution, orally, once daily on Day 1 and Days 4 through 10 (Cohorts 1, 2 and 3), or TAK-058 placebo-matching solution, orally, once on Day 1 (Cohort 5), in non-elderly healthy participants.
  Interventions: Drug: TAK-058 Placebo
- Cohort 4 Elderly Healthy: Placebo (Placebo Comparator): TAK-058 placebo-matching solution, orally, once daily on Day 1 and Days 4 through 10, in non-elderly healthy participants.
  Interventions: Drug: TAK-058 Placebo

INTERVENTIONS:
Drug: TAK-058 — TAK-058 Solution
  Arms: Cohort 1 Non-elderly Healthy: TAK-058 25 mg; Cohort 2 Non-elderly Healthy: TAK-058 75 mg; Cohort 3 Non-elderly Healthy: TAK-058 150 mg; Cohort 4 Elderly Healthy: TAK-058 25 mg; Cohort 5 Non-elderly Healthy: TAK-058 300 mg
Drug: TAK-058 Placebo — TAK-058 placebo-matching solution
  Arms: Cohort 4 Elderly Healthy: Placebo; Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple doses of TAK-058 in healthy non-elderly and elderly participants.

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-058, which is under evaluation for the treatment of schizophrenia.

This study will enroll approximately 32 healthy non-elderly and 8 healthy elderly participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the five treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Cohort 1 Non-elderly Healthy: TAK-058 25 mg
* Cohort 2 Non-elderly Healthy: TAK-058 75 mg
* Cohort 3 Non-elderly Healthy: TAK-058 150 mg
* Cohort 4 Elderly Healthy: TAK-058 25 mg
* Cohort 5 Non-elderly Healthy: TAK-058 300 mg
* Cohort 1-4 Non Elderly Placebo (dummy inactive solution) - this is an oral solution that looks like the study drug but has no active ingredient.
* Cohort 5 Elderly Placebo This single-center trial will be conducted in the United States. The overall time to participate in this study is 40 days if assigned to Cohort 1 to 4. Participants will be confined to the clinic for 12 days, and will be contacted by telephone 11 and 30 days after last dose of study drug for a follow-up assessment (Days 21 and 40).

The overall time to participate in this study is 14 days if assigned to Cohort 5. Participants will be confined to the clinic for 4 days, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment (Day 14).

ELIGIBILITY:
Inclusion Criteria:

* Ages for this study are 18 to 60 years for non-elderly and 18 to 65 years for elderly.
* A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
* A female participant with no childbearing potential, which is defined as the subject has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 years and follicle-stimulating hormone [FSH]>40 IU/L).
* Weighs at least 45 kg (99 lbs) and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive at Screening.

Exclusion Criteria:

* Has received any investigational compound within 30 days prior to the first dose of study medication.
* Has received TAK-058 in a previous clinical study.
* Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
* Has a known hypersensitivity to any component of the formulation of TAK-058.
* Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 6 months prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
* Female participants of childbearing potential (premenopausal, non-sterilized), or has a positive pregnancy test.
* Male participants that intend to donate sperm during the course of this study or for 12 weeks thereafter.
* Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the subject's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-058, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders and cardiac arrhythmias.
* Has previously had a seizure or convulsion (lifetime), including absence seizure and febrile convulsion.
* Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
* Has a history of cancer or other malignancy, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
* Has a positive test result for hepatitis B surface antigen (HBsAg), antibody to hepatitis C virus (anti-HCV) or a known history of human immunodeficiency virus infection at Screening.
* Has poor peripheral venous access.
* Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to Day 1.
* Has a Screening or Check-in (Day -1) abnormal (clinically significant [CS]) electrocardiogram (ECG).
* Has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 60 to 90 mm Hg for diastolic, confirmed with one repeat testing within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1) Visit.
* Has a resting heart rate outside the range 50 to 100 bpm, confirmed with repeat testing within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1) Visit.
* Has a QT interval with Fridericia's correction method (QTcF) >450 ms (males) or >470 ms (females) or PR outside the range of 120 to 220 ms, confirmed with one repeat testing within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1) Visit.
* Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a CS underlying disease or subject with the following lab abnormalities: ALT and/or AST >1.5 the upper limits of normal.
* Has a risk of suicide according to the investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [C-SSRS]) or has made a suicide attempt in the previous 6 months.
* Has uncontrolled, CS neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the subject to participate or potentially confound the study results.
* Has used nicotine-containing products (including but not limited to cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austsitn, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 20 February 2015 to 3 December 2015.
Pre-assignment Details: Healthy non-elderly were enrolled in 1 of 5 treatment groups, TAK-058 25 mg, 75 mg, 150 mg, 300 mg or placebo. Healthy elderly participants were enrolled in 1 of 2 treatment groups, TAK-058 25 mg or placebo.
Groups:
- Cohort 5 Non-elderly Healthy: TAK-058 300 mg: TAK-058 300 mg solution, orally, once on Day 1, in non-elderly healthy participants.
Period: Overall Study
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo
Started | 6 | 6 | 6 | 6 | 6 | 8 | 2
Completed | 6 | 6 | 6 | 6 | 6 | 8 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set, all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (6.77) | 36.2 (11.65) | 42.2 (11.23) | 68.2 (1.83) | 41.0 (15.39) | 40.9 (13.67) | 72.5 (2.12) | 46.6 (15.56)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 2 | 0 | 2 | 12
  Male | 4 | 4 | 4 | 4 | 4 | 8 | 0 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 0 | 3 | 2 | 0 | 1 | 2 | 0 | 8
  White | 5 | 3 | 4 | 5 | 5 | 4 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 2 | 1 | 1 | 3 | 1 | 14
  Not Hispanic or Latino | 1 | 5 | 4 | 5 | 5 | 5 | 1 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 6 | 8 | 2 | 40
Height [Mean (Standard Deviation); unit: cm] | 171.5 (10.17) | 171.0 (7.95) | 173.2 (10.23) | 173.7 (12.21) | 171.0 (9.42) | 176.1 (4.52) | 154.5 (2.12) | 172.0 (9.45)
Weight [Mean (Standard Deviation); unit: kg] | 76.15 (9.291) | 75.63 (10.397) | 83.55 (12.902) | 83.08 (10.778) | 74.17 (15.687) | 79.63 (9.721) | 68.35 (5.869) | 78.23 (11.322)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.87 (1.742) | 25.80 (2.392) | 27.68 (1.451) | 27.48 (1.094) | 25.17 (3.463) | 25.66 (2.942) | 28.60 (1.697) | 26.36 (2.416)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 6 | 6 | 4 | 4 | 5 | 7 | 2 | 34
  Current Smoker | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 6
Caffeine Consumption [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 2 | 5 | 4 | 3 | 1 | 20
  No | 4 | 3 | 4 | 1 | 2 | 5 | 1 | 20
Alcohol Consumption [Count of Participants; unit: Participants]
  Never Drunk | 3 | 5 | 0 | 3 | 4 | 3 | 2 | 20
  Current Drinker | 2 | 0 | 3 | 3 | 2 | 3 | 0 | 13
  Ex-drinker | 1 | 1 | 3 | 0 | 0 | 2 | 0 | 7
Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 5
  Surgically Sterile | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 7
  Female of Childbearing Potential | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Applicable (Participant is Male) | 4 | 4 | 4 | 4 | 4 | 8 | 0 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Cohorts 1-4 Day 1 to Day 40; Cohort 5 Day 1 to Day 14
Population: Safety Set, all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
percentage of participants | 50.0 | 50.0 | 33.3 | 66.7 | 33.3 | 25.0 | 50.0

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post-Dose
Description: The percentage of participants with any markedly abnormal standard safety laboratory values (chemistry and hematology) collected throughout study.
Time Frame: Cohorts 1-4 Day 1 to Day 40; Cohort 5 Day 1 to Day 14
Population: Safety Set, all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 12.5 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Signs at Least Once Post-Dose
Description: The percentage of participants with any markedly abnormal standard vital sign values collected throughout study. Vital signs included blood pressure (after 5 minutes supine and at 1 and 3 minutes after standing), pulse and oral temperature.
Time Frame: Cohorts 1-4 Day 1 to Day 40; Cohort 5 Day 1 to Day 14
Population: Safety Set, all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
percentage of participants
  Any Markedly Abnormal Vital Sign | 16.7 | 66.7 | 50.0 | 50.0 | 50.0 | 12.5 | 100.0
  Pulse Rate | 0.0 | 33.3 | 50.0 | 16.7 | 16.7 | 12.5 | 0.0
  Systolic Blood Pressure | 16.7 | 16.7 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0
  Diastolic Blood Pressure | 16.7 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Temperature | 0.0 | 16.7 | 16.7 | 33.3 | 33.3 | 0.0 | 100.0

4. Secondary Outcome: Mean Cmax: Maximum Observed Plasma Concentration for TAK-058
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 predose and at multiple time points (up to 72 hours) postdose, and Day 10 predose and at multiple time points (up to 24 hours) postdose
Population: Pharmacokinetic Set, all participants who were in the safety set and had at least 1 measurable plasma concentration or amount of drug in urine.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 1076.0 (272.66) | 2085.0 (492.70) | 2366.7 (738.88) | 811.8 (179.48) | 3361.7 (479.85)
  Day 10 | 1035.0 (404.58) | 2021.7 (577.91) | 2158.3 (560.69) | 886.2 (332.50) | NA (NA) — This cohort received a single dose on Day 1 only, therefore Day 10 analysis not applicable.

5. Secondary Outcome: Mean AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-058
Description: AUClast is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration.
Time Frame: Day 1 predose and at multiple time points (up to 72 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 4414.6 (1461.59) | 9223.2 (5433.05) | 12262.6 (4671.88) | 4326.8 (1287.86) | 15143.1 (3471.42)

6. Secondary Outcome: Mean AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-058
Description: AUC24 is measure of area under the curve from time 0 to 24 hours postdose.
Time Frame: Day 1 predose and at multiple time points (up to 24 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 4372.6 (1436.73) | 8862.9 (4782.64) | 12013.0 (4495.56) | 4244.9 (1243.28) | 14852.3 (3348.62)

7. Secondary Outcome: Mean AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-058
Description: Area under the plasma concentration-time curve during a dosing interval, where tau (τ) is the length of the dosing interval.
Time Frame: Day 10 predose and at multiple time points (up to 24 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 4295.3 (2208.92) | 8325.4 (4642.29) | 11905.9 (4447.14) | 4539.2 (1509.66)

ADVERSE EVENTS:
Time Frame: Collection of AEs commenced from the time that the participant was first administered study medication on Day 1 until 30 days following last dose (up to Day 40 for Cohorts 1-4 and up to Day 30 for Cohort 5).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1 Non-elderly Healthy: TAK-058 25 mg | Cohort 2 Non-elderly Healthy: TAK-058 75 mg | Cohort 3 Non-elderly Healthy: TAK-058 150 mg | Cohort 4 Elderly Healthy: TAK-058 25 mg | Cohort 5 Non-elderly Healthy: TAK-058 300 mg | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo | Cohort 4 Elderly Healthy: Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 2/6 | 4/6 | 2/6 | 2/8 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Non-elderly Healthy: TAK-058 25 mg (N=6) | Cohort 2 Non-elderly Healthy: TAK-058 75 mg (N=6) | Cohort 3 Non-elderly Healthy: TAK-058 150 mg (N=6) | Cohort 4 Elderly Healthy: TAK-058 25 mg (N=6) | Cohort 5 Non-elderly Healthy: TAK-058 300 mg (N=6) | Cohorts 1, 2, 3 and 5 Non-elderly Healthy: Placebo (N=8) | Cohort 4 Elderly Healthy: Placebo (N=2)
Infrequent bowel movements (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Application site irritation (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.